CLINICAL TRIAL: NCT03306680
Title: SUNSET: SBRT for Ultra-central NSCLC- a Safety and Efficacy Trial
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUNSET
Record Dates: First submitted 2017-09-28; First posted 2017-10-11 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with ultra-central NSCLC T1-3 (<6cm) N0 M0 (Experimental): Level-1 Dose per fraction: 4Gy Number of fractions: 15 Total Dose: 60 Gy
  Level 0 Dose per fraction: 6Gy Number of fractions: 10 Total Dose: 60 Gy
  Level 1 Dose per fraction: 7.5 Gy Number of fractions: 8 Total Dose: 60 Gy
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Patients will be assigned to treatment doses using the TITE-CRM model.

SUMMARY:
This multi-centre phase I dose-escalation study will use a time-to-event continual reassessment method (TIT-CRM).

Accrual will start at level 1 (60 Gy in 8 fractions). Patients will be assigned to treatment doses using the TITE-CRM model. The model will use all available information from previously accrued patients to assign the highest dose with a predicted risk of grade 3 toxicity of 30% or less.

DETAILED DESCRIPTION:
This study will use a time-to-event continual reassessment method (TITE-CRM). The study design is based on RTOG 0813 (described above), but with a more cautious approach, since the patients herein may constitute a high-risk subset of the patients enrolled in RTOG 0813. The modifications include a starting dose (60 Gy in 8 fractions) herein that is lower than the safe dose for central tumors as determined by RTOG 0813 (60 Gy in 5 fractions), and longer follow-up period during which patients are considered at-risk for toxicity, (i.e. two years herein vs. one year in RTOG 0813).

The primary endpoint of this study is the maximally tolerated dose (MTD) of radiotherapy for ultracentral tumors. The MTD is the dose of radiotherapy associated with a <30% rate of grade 3-5 toxicity occurring within 2 years of treatment.

Local Progression, Regional nodal progression, Distant metastases, Progression-Free Survival, Overall survival, patient reported outcomes and quality of life.

The correlative objectives of this study are to determine the prognostic value of ctDNA levels measured pre-treatment, at the end of treatment and 3- and 12-months after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically (histologically or cytologically) proven diagnosis of non-small cell lung cancer (NSCLC); if the risk of biopsy is unacceptable, pathologic confirmation is not required providing there is serial growth on serial (>=2) CT imaging and/or FDG avidity that is strongly suggestive of a primary NSCLC.
2. Stage T1-3, N0, M0 (UICC/AJCC Staging, 8th Ed.), tumor size < 6 cm, prior to registration, based upon the following minimum diagnostic workup:

   1. History/physical examination within 4 weeks prior to registration
   2. CT scan with contrast (unless medically contraindicated) within 12 weeks of registration. The CT scan will include the entirety of both lungs, the mediastinum, liver and adrenal glands; the primary tumor dimensions will be measured on CT. Note: Patients with lesions that cannot be visualized by CT scan are not eligible for the study.
   3. Whole body positron emission tomography (PET) scan within 12 weeks of registration, using FDG with adequate visualization of the primary tumor and draining lymph node basins in the hilar and mediastinal regions.
   4. Mediastinal lymph node sampling by any technique is encouraged but not required. Patients with hilar or mediastinal lymph nodes <1 cm and no abnormal hilar or mediastinal uptake on PET will be considered N0. Patients with > 1 cm hilar or mediastinal lymph nodes on CT or abnormal PET (including suspicious but nondiagnostic uptake) may still be eligible if directed tissue biopsies of all abnormally identified areas are negative for cancer.
3. ECOG performance status 0-2;
4. age >18;
5. Ultra-central tumor location: tumours whose planning target volume (PTV) is expected to touch or overlaps the central bronchial tree, esophagus, pulmonary vein, or pulmonary artery as determined at the time of consultation.

Exclusion Criteria:

1. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 2 years (e.g. carcinomas in situ of the breast, oral cavity, or cervix are permissible); previous lung cancer, if the patient is disease-free for a minimum of 2 years is permitted.
2. Any prior thoracic radiotherapy.
3. Any prior chemotherapy for the study cancer (cancer proposed to be treated on the study).
4. Prior surgery for the study cancer.
5. Plans for the patient to receive other local therapy (including standard fractionated radiotherapy and/or surgery) while on this study, except at disease progression;
6. Plans for the patient to receive systemic therapy (including standard chemotherapy or biologic targeted agents), while on this study, except at disease progression.
7. Pregnancy.
8. The following autoimmune and connective tissue diseases will be excluded: Scleroderma and Systemic lupus erythematosus
9. patients with interstitial lung disease (ILD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-19 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Maximally tolerated dose (MTD) | Occurring within 2 years of treatment
  MTD of radiotherapy for ultracentral tumors. The MTD is the dose of radiotherapy associated with a <30% rate of grade 3-5 toxicity occurring within 2 years of treatment.

SECONDARY OUTCOMES:
Time to Local Progression | 3-5 years
Regional nodal progression | 3-5 years
  Defined as presence of enlarged lymph nodes >1 cm [short axis] in the hilum or mediastinum.
Time to distant metastases | 3-5 years
Progression-Free Survival | 3-5 years
Overall survival | 3-5 years
Patient reported outcome | Before treatment & at 3, 6, 9, 12, 18, 24, 36, 48, and 60 months
  FACT-L
Quality of Life | Before treatment & at 3, 6, 9, 12, 18, 24, 36, 48, and 60 months
  EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Giuliani, MBBS, FRCPC, Principal Investigator — Princess Margaret Cancer Center
Locations (7):
- Canada (7):
  - BC Cancer -Vancouver Island, Vancouver, British Columbia
  - London Regional Cancer Program, London, Ontario
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - McGill University Health Centre-Cedars Cancer Centre, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rosenberg SA, Mak R, Kotecha R, Loo BW Jr, Senan S. The Nordic-HILUS Trial: Ultracentral Lung Stereotactic Ablative Radiotherapy and a Narrow Therapeutic Window. J Thorac Oncol. 2021 Oct;16(10):e79-e80. doi: 10.1016/j.jtho.2021.06.030. No abstract available. PMID 34561039